CLINICAL TRIAL: NCT04681183
Title: Pilot Study Evaluating Neuro-Imaging Correlates of Epigenetic Finding in Prediction of Chronic Postsurgical Pain
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0277
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Chronic Post-surgical Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be isolated from blood samples and be used for pyrosequencing studies to obtain DNA methylation information for a specified set of genes or use of the Methylation EPIC array.
  DNA samples gathered will be held for future analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This pilot research study is being performed to learn more about pain and look at how pain changes brain chemistry and function. The research team would like to learn new information to better control chronic pain after surgery. This information collected in this research will be used to plan possible future visits. Participants in this study are being asked to participate because they are scheduled for an upcoming surgery. The research team would like to observe them before and after their surgery.

DETAILED DESCRIPTION:
This study is a pilot feasibility study in 30 healthy, preoperative children and young adults undergoing major surgery with high risk for chronic post-surgical pain (CPSP) to characterize the brain metabolite status of the Anterior cingulate cortices (ACC) and insula in pre-surgical adolescents and to understand the relationship between metabolite levels and CPSP. The investigators will also examine whether neurochemical tone in these regions is related to resting state functional connectivity with other brain regions. Correlations between differentially methylated CpG sites in genes enriching gamma aminobutyric acid (GABA) and Dopamine-DARPP-32 pathways and Glu/GABA levels in insula/ACC will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 8 yrs of age
2. English speaking;
3. Healthy (Defined as American Society of Anesthesiologists Physical Status 1 or 2)
4. Ability to provide assent/consent/parent permission.
5. Scheduled to undergo chest surgery (thoracotomy, thoracoscopy, Nuss procedure, pectus surgery, mastectomy), spine surgery, amputation, hernia repair or hip/knee replacement.

Exclusion Criteria:

1. History of chronic pain conditions including migraines
2. Use of opioids chronically or for major surgery within the 6 months prior to enrollment
3. Severe obesity (BMI>35 kg/m2)
4. Taking no more than two concomitant medications known to induce or inhibit CYP2D6 activity, including paroxetine, fluoxetine, cimetidine, and duloxetine or other medications used to treat attention deficit hyperactivity disorder (medications containing amphetamine or methylphenidate).
5. Use of hormonal contraceptives
6. Use of medications that may alter pain sensitivity (e.g. gabapentin,/pregabalin amitryptiline/other antidepressants, clonidine).
7. Active or history of renal/liver problems or congenital cardiac disease
8. Diagnosed developmental delay
9. Pregnant or lactating females
10. Any skin condition that prevents cuff application
11. History of seizures
12. Claustrophobia
13. Metallic implants/orthodontics/braces or other MRI exclusion (MRI safety screening will be conducted prior to enrollment and prior to each MRI scan)

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing chest surgery (thoracotomy, thoracoscopy, Nuss procedure, pectus surgery, mastectomy), spine surgery, amputation, hernia repair or hip/knee replacement in the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Chronic post-surgical pain; Unabbreviated scale title "Chronic post-surgical pain scores" | 2-6 months after surgery
  Pain scores over prior 2 weeks reported 2-6 months after surgery; minimum value = 0, maximum value = 10; higher score means more severe pain

SECONDARY OUTCOMES:
Evoked pressure pain measures; Unabbreviated scale title "Evoked pressure pain measures" | 1-2 weeks after surgery
  Average of 3 measurements taken using a hand-held algometer; minimum value = 0, maximum value = None; higher measurement means better pain tolerance
Resting state connectivity | 1 - 8 weeks before surgery
  Pressure cuff measurements while undergoing MRI scan
Correlation of DNAm of specified gene regions with outcomes | 1-8 weeks before surgery or day of surgery
  Differential DNAm measured by array/sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Vidya Chidambaran, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States